CLINICAL TRIAL: NCT00917865
Title: Anti-[18F]FACBC PET-CT for the Characterization of Primary Prostate Cancer
Brief Title: FACBC Positron Emission Tomography/Computed Tomography(PET/CT) Used in the Diagnosis of Primary Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Optimal histolgic verification support such as whole mount analysis could not be made available.
Sponsor: David M. Schuster, MD (Other)
Responsible Party: Sponsor-Investigator, David M. Schuster, MD, Sponsor-Investigator, Emory University
Organization: Emory University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00008094; FACBC (Other: Other)
Record Dates: First submitted 2009-06-05; First posted 2009-06-10 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2013-11

CONDITIONS: Prostate Cancers
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FACBC Imaging (Experimental): Dynamic FACBC PET of primary prostate carcinoma.
  Interventions: Drug: anti [18F]FACBC

INTERVENTIONS:
Drug: anti [18F]FACBC — Anti[18F]FACBC (10mci) will be given intravenously over 1-2 minutes prior to obtaining PET-CT images At 4 minutes, 10 consecutive/4minutes images will be obtained of the pelvis to include the prostate.

SUMMARY:
The purpose of this research project is to test if a compound (chemical substance) has a natural tendency to go to prostate cancer. This compound has a small amount of radioactivity attached to it and is called a radiotracer. The name of the radiotracer is FACBC and can be detected on a special imaging device called a PET scanner (positron emission tomography). The radiotracer is treated in the body much like an amino acid which is a nutrient required for normal functioning. Tumors also use these nutrients. Earlier studies have shown that this radiotracer may be able to detect prostate cancer.

The investigators will perform a study with 20 patients in whom they know have prostate cancer after a biopsy and who are scheduled for an operation in which the prostate is removed and the nearby lymph nodes are examined. This operation is called prostatectomy. The investigators think that this radiotracer can help us determine where exactly the prostate cancer is present in the prostate or if it has spread. This information may be useful in the future to help with other non-surgical therapy such as radiation beam therapy.

The investigators will compare the results of the FACBC PET scan to the results of the pathology analysis of the removed prostate. In this way the investigators can determine how good a test FACBC PET is for finding out where and if prostate cancer is located in the prostate or nearby lymph nodes. The investigators will also do more advanced analysis on the biopsy samples to see if they can tell why FACBC goes into prostate cancer cells.

This radiotracer has been tested in over 100 human subjects without incident. It has also been chosen by the National Institutes of Health (NIH) as a promising radiotracer. The NIH is funding this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older.
* Patients will be scheduled for prostatectomy based on a diagnosis of primary prostate cancer.
* Ability to lie still for PET scanning
* Patients must be able to provide written informed consent.

Exclusion Criteria:

* Age less than 18
* Inability to lie still for PET scanning
* Cannot provide written informed consent.
* Less than 4 weeks since any prior prostate biopsy (to decrease false positive uptake from inflammation).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Schuster, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Schuster DM, Taleghani PA, Nieh PT, Master VA, Amzat R, Savir-Baruch B, Halkar RK, Fox T, Osunkoya AO, Moreno CS, Nye JA, Yu W, Fei B, Wang Z, Chen Z, Goodman MM. Characterization of primary prostate carcinoma by anti-1-amino-2-[(18)F] -fluorocyclobutane-1-carboxylic acid (anti-3-[(18)F] FACBC) uptake. Am J Nucl Med Mol Imaging. 2013;3(1):85-96. Epub 2013 Jan 5. PMID 23342303
- See also: Click here for more information on this study — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3545368/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 5/2008-3/2011. Subjects were referred from physician's offices
Groups:
- Radiotracer: [18F] FACBC 10mci injected intravenously prior to PET scan
Period: Overall Study
Arm/Group | Radiotracer
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiotracer
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 60.8 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Performance Per Sextant at Each Time Point by Visual Analysis
Description: Each of 12 sextants per prostate (for a total of 120 sextants for the 10 patients) were analyzed separately at 4, 16, 28 and 40 min post-injection for the presence or absence of focal activity suspicious for tumor.
  Sensitivity: Proportion of people with a disease who have a positive test result
  Specificity: The proportion of people without disease who have a negative test result Positive Predictive Value (PPV):The probability that a person who has a positive test result has the disease for which the test was conducted.
  Negative Predictive Value (NPV): The probability that a person who has a negative test result does not have the disease for which the test was conducted
  Accuracy: Ability of the test to differentiate between disease and non-disease.
  Note: 'n=' is the denominator used to compute each parameter.
Time Frame: At 4, 16, 28 and 40 minutes post-injection of FACBC
Population: The number of participants for analysis was based on the protocol.Each prostate was divided into 12 sextants and then each sextant was visualized for abnormal focal uptake.The SUVmax for the malignant sextants were compared to that of the benign sextants. Note: 'n=' is the denominator used to compute each parameter.
Measure: Number (95% Confidence Interval); unit: Percentage of Sextants
Units Other Than Participants: Sextants
Groups:
- Diagnostic Performance Per Sextant at 4mins Post Injection: Each of the 120 sextants was visually analyzed for the presence or absence of tumor. 71 true positive, 7 True negative, 32 false positive and 8 false negative. Because of a technical error, 2 of the 120 sextants were not analysed at this time point.
- Diagnostic Performance Per sextant16mins Post Injetion: At this time point, the 120 sextants analysed were categorized as followed:
  68 sextants were seen as true positive, 14 true negative, 25 false positive and 13 false negative
- Diagnostic Performance Per Sextant 28mins Post Injection: At this time point, the 120 sextants analysed were categorized as followed:
  65 sextants were seen as true positive, 20 true negative, 20 false positive and 15 false negative
- Diagnostic Performance Per Sextant 40minutes Post Injection: At this time point, the 120 sextants analysed were categorized as followed:
  63 sextants were seen as true positive, 15 true negative, 25 false positive and 17 false negative
Arm/Group | Diagnostic Performance Per Sextant at 4mins Post Injection | Diagnostic Performance Per sextant16mins Post Injetion | Diagnostic Performance Per Sextant 28mins Post Injection | Diagnostic Performance Per Sextant 40minutes Post Injection
Number analyzed (Participants) | 10 | 10 | 10 | 10
Number analyzed (Sextants) | 118 | 120 | 120 | 120
Percentage of Sextants
  Sensitivity (n=79, 81, 80, 80) | 89.9 (2.6) [80.5 to 95.2] | 84.0 (1.6) [73.8 to 90.9] | 81.3 (1.3) [70.6 to 88.8] | 78.8 (1.0) [67.9 to 86.8]
  Specificity (n = 39, 39, 40, 40) | 18.0 [8.1 to 34.1] | 35.9 [21.7 to 52.9] | 50.0 [34.1 to 65.9] | 37.5 [23.2 to 54.2]
  PPV (n = 103, 93, 85, 88) | 68.9 [59.0 to 77.5] | 73.1 [62.8 to 81.5] | 76.5 [65.8 to 84.7] | 71.6 [60.8 to 80.5]
  NPV (n = 15, 27, 35, 32) | 46.7 [22.3 to 72.6] | 51.9 [32.4 to 70.9] | 57.1 [39.5 to 73.2] | 46.9 [29.5 to 65.0]
  Accuracy (n = 118, 120, 120, 120) | 66.1 [56.7 to 74.4] | 68.3 [59.1 to 76.4] | 70.8 [61.7 to 78.6] | 65.0 [55.7 to 73.3]

2. Secondary Outcome: Mean SUVmax of Low Versus High Gleason Groups
Description: To determine id radiotracer uptake correlates with gleason score
Time Frame: 4 minutes,16 minutes,28 minutes and 40 minutes
Measure: Mean (Standard Deviation); unit: Mean SUV max
Groups:
- Mean SUV Max at 4 Minutes: The 79 malignant sextants were grouped according to their Gleason score. Low Gleason: 3+3 and 3+4 High Gleason: 4+3, 4+4, 5+5 The SUV max was then determined for each group at 4 minutes
- Mean SUV Maxat 16 Minutes: The 79 malignant sextants were grouped according to their Gleason score. Low Gleason: 3+3 and 3+4 High Gleason: 4+3, 4+4, 5+5 The SUV max was then determined for each group at 16 minutes
- Mean SUV Max at 28 Minutes: The 79 malignant sextants were grouped according to their Gleason score. Low Gleason: 3+3 and 3+4 High Gleason: 4+3, 4+4, 5+5 The SUV max was then determined for each group at 28 minutes
- Mean SUV Maxat 40minutes: The 79 malignant sextants were grouped according to their Gleason score. Low Gleason: 3+3 and 3+4 High Gleason: 4+3, 4+4, 5+5 The SUV max was then determined for each group at 40 minutes
Arm/Group | Mean SUV Max at 4 Minutes | Mean SUV Maxat 16 Minutes | Mean SUV Max at 28 Minutes | Mean SUV Maxat 40minutes
Number analyzed (Participants) | 10 | 10 | 10 | 10
Mean SUV max
  Low gleason group | 4.4 (2.1) | 3.8 (1.1) | 3.5 (1.0) | 3.3 (0.9)
  High gleason group | 5.9 (2.8) | 5.2 (1.7) | 4.7 (1.3) | 3.3 (0.9)

ADVERSE EVENTS:
Arm/Group | Radiotracer
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
A major limitation of our study is lack of step section whole mount histology at our institution which restricted the ability to ensure an exact correlation of histology to imaging.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No